CLINICAL TRIAL: NCT05437367
Title: Effect of Scapular Stabilization Exercises on Scapular Muscles Strength and Kyphosis Index in Smartphone Users
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Soliman Mohamed Soliman, Principal investigator, Cairo University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: P.T.REC/012/003673
Record Dates: First submitted 2022-06-18; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Muscle Weakness; Smartphone Addiction
MeSH Terms: conditions — Muscle Weakness; Internet Addiction Disorder

STUDY DESIGN:
Intervention Model Description: Randomized experimental, controlled study (pretest- posttest measurement). Inclusion Criteria
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- posture correction exercises group 1 (Other): Group A (Control group 1): Participants using smartphones more than 4 hours per day will receive posture correction exercises only.
  Interventions: Other: Postural correction exercises
- scapular stabilization and postural correction exercises group 1 (Experimental): Group B (Experimental group 1): Participants using smartphones more than 4 hours per day will receive scapular stabilization and postural correction exercises.
  Interventions: Other: Scapular Stabilization exercises; Other: Postural correction exercises
- posture correction exercises group 2 (Other): Group C (Control group 2): Participants using smartphones less than 4 hours per day will receive posture correction exercises only.
  Interventions: Other: Postural correction exercises
- scapular stabilization and postural correction exercises group 2 (Experimental): Group D (Experimental group 2): Participants using smartphones less than 4 hours per day will receive scapular stabilization and postural correction exercises.
  Interventions: Other: Scapular Stabilization exercises; Other: Postural correction exercises

INTERVENTIONS:
Other: Scapular Stabilization exercises — Therapeutic exercises
  Arms: scapular stabilization and postural correction exercises group 1; scapular stabilization and postural correction exercises group 2
Other: Postural correction exercises — Therapeutic exercises

SUMMARY:
This study will be conducted to investigate the effect of scapular stabilization exercises on scapular muscles strength (serratus anterior, lower fibers of trapezius, rhomboid major and minor), pain intensity level and kyphosis index in different duration of time using daily of smartphone in smartphone users.

DETAILED DESCRIPTION:
Modern people use a smartphone along the day, including occupational and leisure activities. Repeated and prolonged use of smartphones affecting muscular activity and strength around the shoulders and upper back especially serratus anterior during maintaining an un ideal posture which may result in the development of postural changes as excessive thoracic kyphosis which in turn will result in inadequate muscles contractions, weakening of postural muscles and fatigue. Scapular muscles strength should be balanced or integrated (muscle balance) and worked in synchronized motion, so, alteration in scapulothoracic motion in resting position or dynamic motion of scapula described as scapulothoracic dysfunction. Muscle imbalances occurs and lower trapezius, serratus anterior and rhomboids muscles are the most common muscles prone to weakness due to exposure to sustained awkward posture or adaptive postures and restriction to specific activity. Continuous use of smartphone for more than 4 hours daily increases shoulder and parascapular pain, fatigue, decrease strength of scapular muscles (lower fibers of trapezius for scapular adduction and depression and rhomboids for scapular adduction and downward rotation) in right dominant side due to prolonged hyperactivity, then weakness.The excessive use of smartphones correlates with increases incidence of vertebral static disorders, especially kyphosis.

Scapular stabilization exercises were effective in the early rehabilitation and the balance of both sides of the trapezius with the movement and couple motion of the scapula. It is also effective in increasing muscle activation in the serratus anterior and lower trapezius.

ELIGIBILITY:
Inclusion Critria

* Normal subjects from both genders.
* Subjects had to be right hand dominant.
* Age ranged from 17 to 45 years old.
* All subjects had at least 6 months experience in using touch-screen smartphones.
* The mean of smartphone size included in the study will be 5 inches (Mohamed et al., 2020).

Exclusion Criteria:

* Any pain or limitation (dysfunction) at neck and shoulder.
* Any congenital abnormalities in either the cervical or the lumbar spine.
* Previous history of severe surgical procedures.
* Any history of upper extremity injury within the past year.
* Visual problems, dizziness and vertigo.
* Any deformity in the upper extremities or spine.
* Neurological or systemic disorders.
* If they had taken any sedative drug or alcohol within the past 48 hours.

Ages: 17 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 88 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of change in scapular Muscles strength | at baseline and after 4 weeks of intervention
  To assess the change in scapular Muscles strength by pull push dynamometer (Newton).
Assessment of change in kyphosis Index | at baseline and after 4 weeks of intervention
  To assess the change in kyphosis Index for thoracic spine pre and post scapular Stabilization exercises for smartphone users by flexible ruler.
Assessment of change in pain intensity level | at baseline and after 4 weeks of intervention
  To assess the change in pain intensity level using visual analog scale (scores) (score 0: means no pain & score 10: means highest pain)

CONTACTS AND LOCATIONS:
Overall Officials: Amira Hussin, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Dokki, Outpatient Clinic, Faculty of Physical Therapy, Egypt